CLINICAL TRIAL: NCT01157728
Title: Early Cognitive Impairment in Multiple Sclerosis: a Multimodal MRI Study Evaluating the Relative Contribution of Cortical and White Matter Tract Injury
Brief Title: Early Cognitive Impairment in Multiple Sclerosis
Acronym: CogniSEP
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: ARSEP (Association pour la Recherche sur la Sclerose en Plaques) (Unknown); JNLF (Journées de Neurologie de Langue Française) (Unknown)
Responsible Party: Sponsor
Other Study IDs: P071102
Record Dates: First submitted 2010-07-06; First posted 2010-07-07 (Estimated); Last update posted 2012-07-31 (Estimated); Status verified 2010-05

CONDITIONS: Multiple Sclerosis; Cognitive Impairment
Keywords: Multiple sclerosis; Cognitive impairment
MeSH Terms: conditions — Multiple Sclerosis; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Relapsing Multiple Sclerosis patients
- healthy volunteer

SUMMARY:
Cognitive impairment is one of the symptoms of Multiple Sclerosis (MS), and it may occur during the first years of the disease. It usually affects attention, information processing speed and short term memory. To date, the mechanisms of this specific symptom remain unclear (local or global inflammation, neurodegenerative processes).

Magnetic Resonance Imaging (MRI) can be useful to understand the pathophysiology of cognitive impairment in MS. The investigators will combine conventional and non conventional MRI sequences to determine the respective role of white matter and grey matter injury and the cortical reorganization of neuronal networks.

DETAILED DESCRIPTION:
Cognitive impairment in Multiple Sclerosis (MS) occurs in 50% of patients and has a major social impact. There is no clear correlation between cognitive dysfunction and disease duration and recent studies have pointed out that it may affects patients at the very early stages of the disease especially in tasks involving sustained attention, processing speed, working memory and executive function.

Recent imaging and pathology studies have shown that MS affects white matter as well as grey matter. Unlike white matter lesion burden or distribution, grey matter atrophy has often been linked to cognitive impairment. Microscopic injury of Normally Appearing White Matter (NAWM) explored by non conventional MRI sequences has also been shown to be involved in pathophysiology of cognitive disorders.

Nevertheless mechanisms of cognitive impairment remain unclear. The relationship between cortical injury and diffuse white matter tracts damage and their respective contribution to cognitive dysfunction affecting patients during the first years of the disease is still under investigation.

This study aims at investigating structural and functional correlates of early cognitive impairment using multimodal MRI.

Relapsing Remitting MS (RRMS) patients with disease duration of less than 5 years will be included. Patients with and without cognitive impairment will be compared to healthy controls. All subjects will perform a clinical and neuropsychological evaluation before the MRI examination.

We will combine new available MRI techniques using a 3 Tesla magnet in order to evaluate precisely cortical and white matter tracts lesions in patients with cognitive MS. These techniques will include :

* 3D T1 sequences to study cortical atrophy using VBM.
* Diffusion tensor imaging fibre tracking to study selected white matter tracts that may be involved in cognitive disorders, such as the thalamus-cortical or the striatum-cortical tracts connecting sub-cortical structures to the prefrontal cortex.
* Functional MRI sequences during a working memory task and during the resting state in order to describe functional networks and their possible reorganization in patients with or without cognitive impairment.

ELIGIBILITY:
Inclusion Criteria:

* Relapsing remitting Multiple Sclerosis patients
* Age: 18-40 years
* Evolving between 3 and 5 years
* EDSS<5

Exclusion Criteria:

* MRI exclusion criteria (metallic prothetic, pace maker etc)
* Renal failure due to Gadolinium injection
* Major depressive disorder

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: * Relapsing remitting Multiple Sclerosis patients
  * Age: 18-40 years
  * Evolving between 3 and 5 years
  * EDSS<5
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2008-05; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Stankoff, MD,PhD, Principal Investigator — Pitié-Salpêtrière Hospital
Locations (1):
- Pitie salpêtrière Hospital, Paris, France